CLINICAL TRIAL: NCT04074343
Title: A Phase Ib Multicenter Study of TAS-102 in Combination With Irinotecan in Patients With Advanced Recurrent or Unresectable Gastric and Gastroesophageal Adenocarcinoma After at Least One Line of Treatment With a Fluoropyrimidine and Platinum Containing Regimen
Brief Title: TAS-102 and Irinotecan in 2L+ Gastric and Gastroesophageal Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Farshid Dayyani, Associate Clinical Professor of Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 18-125 [HS# 2019-5179]; 2019-5179 (Other: University of California, Irvine)
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Gastric Adenocarcinoma; GastroEsophageal Cancer
Keywords: Gastric Adenocarcinoma; TAS-102; Irinotecan; Gastroesophageal Adenocarcinoma
MeSH Terms: interventions — trifluridine tipiracil drug combination; Trifluridine; tipiracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAS-102 and Irinotecan (Experimental): Patients receive TAS-102 25 mg/m2 PO twice daily on days 1-5 and and Irinotecan 180mg/m2 IV on day 1 every 14 days.
  Interventions: Drug: TAS-102; Drug: Irinotecan

INTERVENTIONS:
Drug: TAS-102 — Given PO
  Other Names: LONSURF; trifluoridine and tipiracil
Drug: Irinotecan — Given IV
  Other Names: CAMPTOSAR; CPT-11

SUMMARY:
This is a phase Ib single-arm, open-label clinical trial determining the feasibility and efficacy of TAS-102 and irinotecan in subjects with advanced gastric and gastroesophageal adenocarcinoma. These are subjects who are not candidates for curative treatments and who have received at least one prior line of chemotherapy with a fluoropyrimidine and platinum agent.

DETAILED DESCRIPTION:
Treatment on study will be administered in 14 day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed gastric or gastroesophageal adenocarcinoma
* Must have locally advanced, recurrent, or metastatic disease not amenable to curative intent surgery.
* Must have progressed, or not tolerated, at least one line of treatment with a platinum and/or fluoropyrimidine containing regimen. At least one cycle of combination chemotherapy including a platinum (oxaliplatin, cisplatin, carboplatin) and/or fluoropyrimidine (capecitabine or 5-Fluorouracil) based regimen for advanced disease. Combination regimens with platinum/fluoropyrimidine containing a taxane and or a checkpoint inhibitor are allowed. Patients progressing within six months of perioperative chemotherapy or definitive chemoradiation for localized disease are eligible. Patients who have exhausted all other standard of care options are also eligible.
* Age ≥ 18 years
* Performance status: ECOG performance status ≤2
* Life expectancy of greater than 3 months
* Adequate organ and marrow function as defined below:

  1. leukocytes : ≥ 3,000/mcL
  2. absolute neutrophil count: ≥ 1,500/mcL
  3. platelets: ≥ 80,000/mcl
  4. total bilirubin: within normal institutional limits
  5. AST(SGOT)/ALT(SPGT): ≤ 3 X institutional upper limit of normal or ≤ 5 X if liver metastases are present
  6. creatinine: < 1.5 X upper limit of normal
* The effects of TAS-102 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because topoisomerase inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  1. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  1. Has not undergone a hysterectomy or bilateral oophorectomy; or
  2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to swallow tablets
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients who have had major surgery within 4 weeks, or chemotherapy or radiotherapy within 2 weeks prior to Cycle 1 Day 1.
* All toxicities attributed to prior anti-cancer therapy other than alopecia must have resolved to grade 1 or baseline
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases due to poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102, irinotecan or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior treatment with irinotecan or TAS-102
* History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ.
* Inability to comply with study and follow-up procedures as judged by the Investigator
* Patients who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Dayyani, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAS-102 and Irinotecan
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 23 patients were screened. Three patients were not eligible, and thus 20 eligible patients started the study treatment.
Arm/Group | TAS-102 and Irinotecan
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 61 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  Hispanic | 6
  Asian | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival at 6 Months
Description: This is defined as the percentage of subjects who are free of progression 6 months after study treatment start. Progression is defined as death, radiographic progression or clinical deterioration attributed to disease progression as judged by an investigator. Radiographic progression is defined using the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of diameters of target lesions and an absolute increase of an least 5 mm and/or appearance of new lesions.
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | TAS-102 and Irinotecan
Number analyzed (Participants) | 20
percent of participants | 40 [19.3 to 60.0]

2. Secondary Outcome: Number of Participants With Grade 3-5 Adverse Events
Description: To evaluate the tolerability of administering TAS-102 in combination with Irinotecan in patients with advanced recurrent or unresectable gastric and gastroesophageal adenocarcinoma for the first 2 cycles of study treatment. Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-102 and Irinotecan
Number analyzed (Participants) | 20
Participants | 8

3. Secondary Outcome: Objective Response Rate as Assessed by RECIST v1.1 Criteria of Patients Who Received TAS-102 and Irinotecan
Description: To assess the objective response rate to the combination of TAS-102 and Irinotecan. Objective response rate (ORR) is defined as confirmed complete response (CR) and partial response (PR). Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. ORR = CR + PR
Time Frame: From date of registration until first date of disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-102 and Irinotecan
Number analyzed (Participants) | 17
Participants | 0

4. Secondary Outcome: Overall Survival of Patients of Patients Who Received TAS-102 and Irinotecan
Description: To evaluate overall survival in patients with advanced recurrent or unresectable and gastroesophageal adenocarcinoma treated with this combination of TAS-102 and Irinotecan.
Time Frame: From date of registration for up to 18 months after last patient is enrolled or until death from any cause, whichever came first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-102 and Irinotecan
Number analyzed (Participants) | 20
Months | 12.2 [5.9 to 18.6]

ADVERSE EVENTS:
Time Frame: From date of registration until treatment completion, disease progression or other reasons for removal from protocol treatments, whichever came first, an average of 1 year.
Description: Toxicity was graded according to National Cancer Institute Common Terminology Criteria of Adverse Events, version 5.0. Safety was assessed through adverse event monitoring, physical examinations, vital signs and clinical laboratory tests before each dosing.
Arm/Group | TAS-102 and Irinotecan
All-Cause Mortality (participants affected / at risk) | 17/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-102 and Irinotecan (N=20)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-102 and Irinotecan (N=20)
Nausea (General disorders) | 14
Diarrhea (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 10
Abdominal Pain (General disorders) | 7
Vomiting (General disorders) | 6
Anorexia (Nervous system disorders) | 6
Alopecia (Immune system disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Headache (General disorders) | 3
Mucositis oral (General disorders) | 2
Hypotention (Vascular disorders) | 2
Neutrophil count decreased (Blood and lymphatic system disorders) | 6
Anemia (Blood and lymphatic system disorders) | 5
Hypokalemia (Blood and lymphatic system disorders) | 2
White blood cell decreased (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT04074343/Prot_SAP_000.pdf